CLINICAL TRIAL: NCT02481804
Title: Towards Optimal Personalized Diet and Vitamin Supplementation in NET Patients; a Pilot Study
Brief Title: Optimal Feeding for NET Patients
Acronym: DIVIT-pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05012015
Record Dates: First submitted 2015-01-06; First posted 2015-06-25 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Neuroendocrine Tumor
Keywords: diet; vitamin
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary intervention (Experimental): There is one arm. Patients will first have an observation period, whre hey will get standard treatment during four weeks. Thereafter they will have the dietary intervention during 14 weeks.
  Interventions: Other: Dietary intervention; Other: Standard treatment

INTERVENTIONS:
Other: Dietary intervention — Patients will be counseled by a dietician for 14 weeks. A tailored diet advice for each NET patient will be based on the individual situation which includes gastrointestinal complaints, the location of the tumor, additional treatments like previous surgery and measured vitamine and tryptophan levels.
  Dietician consults will be conducted by 1 out-patient visit and 3 follow up contacts.
Other: Standard treatment — Standard treatment will be continued

SUMMARY:
This study aims to investigate if optimal personalized consultation by a dietician for a healthy diet focused on food which contains sufficient vitamins and minerals improves gastrointestinal symptoms as determined by an improved score in the gastrointestinal symptoms of the NET specific EORTC QLQ-GINET21 at end of study.

DETAILED DESCRIPTION:
Rationale: Patients with neuroendocrine tumors (NET) have a rare, slowly progressing disease. Therefore they undergo many treatments such as surgery followed by long-lasting systemic treatments with somatostatin analogues. These procedures can each result in increased diarrhea and loss of critical food components in the stools such as fat. This can lead amongst others, to major loss of fat-soluble vitamins. Those patients who in addition have an ongoing serotonin production may experience shortage in the circulating essential amino acid tryptophan. Serotonin is derived from the essential amino acid tryptophan. Tryptophan is a precursor of niacin (vitamin B3) which is critical for normal cellular metabolism. In case of high serotonin production in neuroendocrine tumor patients tryptophan and/or niacin can be deficient leading to symptoms including pellagra. Suppletion of tryptophan might facilitate serotonin production and therefore, is undesirable in patients with serotonin producing neuroendocrine tumors.

Strikingly little is known about how NET patients should be best supported for the deficits they develop during their long-lasting disease. Also the precise effect of diet advices for diarrhea and fat-soluble vitamins and vitamin B3, in this patient group is unknown.

Patients with NET are faced with a serious chronic disease. This makes this patients group extremely motivated to be involved in their treatment and to "self-manage" their disease as much as possible.

Objective: This study aims to investigate if optimal personalized consultation by a dietician for a healthy diet focused on food which contains sufficient vitamins and minerals improves gastrointestinal symptoms as determined by an improved score in the gastrointestinal symptoms of the NET specific EORTC QLQ-GINET21 at end of study. Secondary aims are decrease in distress on the distress thermometer, improvement in quality of life as determined by the cancer-specific EORTC QLQ-C30, and the other constructs of the EORTC QLQ-GINET21, empowerment (subscales of the Construct Empowering Outcomes questionnaire) at end of study, an improvement in nutrition state (Patient-Generated Subjective Global Assessment PG/SGA) and normalization of vitamins and tryptophan levels at end of study measured with quantitative analysis of blood and urine.

Study design: This is a single center 18 week open-label, non-comparative, single-arm, experimental pilot study. In this pilot we want to examine the effect sizes of the gastrointestinal symptoms of the NET specific EORTC QLQ-GINET21 of the patients after the dietary intervention. Four weeks after inclusion adult patients with metastasized NET and chronic use (>6 months) of a somatostatin analogue will start with the dietary intervention. Effects of the intervention will be evaluated by questionnaires and vitamin values in blood and urine.

Patients fill out these questionnaires at baseline, after four weeks, and after 18 weeks. Furthermore at baseline, after four weeks, and after 18 weeks vitamin values in blood and urine will be measured and at baseline.

Study population: Patients that are treated in the University Medical Center Groningen for metastasized NET treated with a somatostatin analogue for more than 6 months will be eligible.

ELIGIBILITY:
Inclusion Criteria:

* Adult NET patients (aged ≥ 18 years of age), with serotonine producing or non-serotonin producing tumors, with any tumor site and disease stage.
* Use of somatostatin analogue for > 6 months.
* Ability to comprehend Dutch (both reading and writing).
* Written informed consent provided.

Exclusion Criteria:

* Estimated life expectancy less than 3 months.
* Patients who have a history of another primary malignancy, except for radical and adequately treated malignancies from which the patient has been disease free for ≥ 3 years.
* Major abdominal surgery during study period.
* Known hypersensitivity of (components of) somatostatin analogue.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
gastro-intestinal symptoms | 18 weeks
  Primary endpoint is the difference in mean gastro-intestinal symptoms score of the EORTC QLQ-GINET21

SECONDARY OUTCOMES:
distress | 18 weeks
  change in distress, as measuerd by the distress thermometer,
quality of life | 18 weeks
  quality of life as determined by the cancer-specific EORTC QLQ-C30, and the other constructs of the EORTC QLQ-GINET21
empowerment at end of study | 18 weeks
  empowerment (subscales of the Construct Empowering Outcomes (CEO) questionnaire) at end of study
nutrition state | 18 weeks
  the difference in the difference in nutrition state (Patient-Generated Subjective Global Assessment PG/SGA)
vitamins and tryptophan levels | 18 weeks
  normalization of vitamins and tryptophan levels at end of study measured with quantitative analysis of blood and urine

CONTACTS AND LOCATIONS:
Overall Officials: A. M.E. Walenkamp, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands